CLINICAL TRIAL: NCT04452448
Title: Analysis of I-Trace High Order Aberrations Induced by Wavefront Optimized Ablation Profiles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030490
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Intervention Model Description: A prospective clinical study including 20 eyes of 10 cases undergoing LASIK with wave front optimized ablation profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser in situ keratomileusis (Experimental): A prospective clinical study including 20 eyes of 10 cases undergoing laser in situ keratomileusis (LASIK)
  Interventions: Device: LASIK

INTERVENTIONS:
Device: LASIK — All cases were operated upon using Wavelight Allegretto EX-500 excimer laser (Alcon Laboratories, Inc., Fort Worth, TX) with wave front optimized ablation profile WFO. The Moria II microkeratome (Moria, Anthony, France) was used in all cases.

SUMMARY:
This work aims at the analysis of ocular aberrations induced by wave front optimized ablation profiles WFO using I-Trace aberrometer (Ray -Tracing)

DETAILED DESCRIPTION:
The iTrace (Tracey Technologies, Houston, Tx) is uniquely designed to combine Placido corneal topography with a ray tracing aberrometer to measure quality of vision in a patient. This work aims at the analysis of ocular aberrations induced by wave front optimized ablation profiles WFO using I-Trace aberrometer (Ray -Tracing)

ELIGIBILITY:
Inclusion Criteria:

1. Myopia up to -8.0 D and astigmatism up to -2.0D.
2. Cases above 18 years of age with a stable refraction for at least one year.

Exclusion Criteria:

1. Keratoconus.
2. Patients with collagen diseases.
3. Previous LASIK or any other refractive surgery.
4. Severe dry eye syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of ocular aberrations | 3 months
  3. Evaluation of ocular aberrations done using iTrace Visual Functional Analyzer (ray tracing technology) to quantify changes in total higher order aberrations, coma, spherical aberrations, secondary astigmatism and trefoil after LASIK surgery
Visual acuity | 3 months
  Unaided as well as best corrected visual acuity
Manifest refraction | 3 months
  Manifest refraction

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mossallam, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No